CLINICAL TRIAL: NCT00742599
Title: Phase III Controlled Clinical Study of NPO-11 in Patients Undergoing Gastric Endoscopy (Randomized, Double-blind, Parallel-assignment , Placebo-controlled Study)
Brief Title: Phase III Controlled Clinical Study of NPO-11 in Patients Undergoing Gastric Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Yasumasa Ogawa, Nihon Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPO-11-01/C-01
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Patients Undergoing Gastric Endoscopy
Keywords: Stomach Diseases
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N (Active Comparator)
  Interventions: Drug: NPO-11
- P (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPO-11 — 20 ml NPO-11
  Arms: N
Drug: Placebo — 20 ml NPO-11(Placebo)
  Arms: P

SUMMARY:
Patients who require gastric endoscopy will receive an intragastric single dose of NPO-11 20 mL. The superiority of NPO-11 to placebo as a premedication for endoscopy will be verified in a randomized, double-blind, parallel-assignment design based on the percentage of patients having no gastric peristalsis at both 2 minutes post-dose and the end of endoscopy (primary outcome measure).

The safety of NPO-11 will be evaluated based on adverse events and adverse drug reactions (ADRs) observed between administration and seven days after administration in comparison with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

Inpatients or outpatients of either sex who visit medical institutions for treatment or follow-up of confirmed or suspected upper gastrointestinal disease (symptoms) and meet the criteria (1) and (2) below will be enrolled in the study. Patients have to provide written informed consent for voluntary participation in the study.

1. Patients who need gastric endoscopy (except for endoscopy with a scope of <9 mm in diameter, emergency endoscopy and endoscopy for comprehensive medical examination)
2. Patients who are older than 20 years at the time of consent

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study. The criteria (2) to (5) will be confirmed during endoscopy. Patients who meet any of these criteria will be withdrawn from the study at the time of confirmation.

1. Patients with a history of surgery to the upper gastrointestinal tract
2. Patients with severe gastric stenosis or deformation which makes observation of gastric peristalsis difficult
3. Patients with upper gastrointestinal bleeding which requires hemostasis
4. Patients with reflux esophagitis (Los Angeles classification: B, C or D)
5. Patients with gastric or duodenal ulcers in active stage
6. Patients on cancer treatment (chemotherapy or radiotherapy)
7. Patients with impaired cardiac function (NYHA functional classification: III or IV)
8. Patients with a history of shock or hypersensitivity to l-menthol or peppermint oil (mint oil)
9. Patients with a history of shock or hypersensitivity to lidocaine hydrochloride
10. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
11. Patients who have been exposed to NPO-11
12. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
13. Patients otherwise ineligible for participation in the study in the investigator's or subinvestigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Presence or absence of gastric peristalsis (central evaluation by independent evaluator) No gastric peristalsis is defined as when patients have no gastric peristalsis at both 2 minutes post-dose and the end of endoscopy. | each evaluation point

SECONDARY OUTCOMES:
Change in gastric peristalsis | each evaluation point
Difficulty level of intragastric observation (evaluation by investigator who performs endoscopy) | each evaluation point
Adverse events and ADRs observed between administration and 7±3 days after administration | each evaluation point

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Kansai
  - Kanto

REFERENCES:
- [Derived] Hiki N, Kaminishi M, Yasuda K, Uedo N, Honjo H, Matsuhashi N, Hiratsuka T, Sekine C, Nomura S, Yahagi N, Tajiri H, Suzuki H. Antiperistaltic effect and safety of L-menthol sprayed on the gastric mucosa for upper GI endoscopy: a phase III, multicenter, randomized, double-blind, placebo-controlled study. Gastrointest Endosc. 2011 May;73(5):932-41. doi: 10.1016/j.gie.2010.12.013. Epub 2011 Feb 26. PMID 21353674